CLINICAL TRIAL: NCT04733846
Title: Treatment of Corneal Wounds Emergencies During the COVID-19 Shutdown: Absorbable 10-0 Vicryl Sutures as a Valuable Strategy.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN202021/CHUSTE
Record Dates: First submitted 2021-02-01; First posted 2021-02-02 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-01

CONDITIONS: Eye Trauma
Keywords: Corneal; penetrating injury; lamellar laceration; COVID; polyglactin; Vicryl
MeSH Terms: conditions — Eye Injuries; Wounds, Penetrating | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- corneal trauma sutured with Vicryl 10-0 monofilament: corneal trauma sutured with Vicryl 10-0 monofilament will be included. They will have data collection of medical records.
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Collection of clinical and paraclinical data during preoperative consultation Collection of clinical and paraclinical data during post-operative consultations Tele-consultation to determine if criteria for good healing / adherence, treatment tolerance / response to questions Remote follow-up 6 and 12 months after the trauma

SUMMARY:
Vicryl (polyglactin) 10-0 resorbable suture is rarely used, little known to ophthalmologists but may offer therapeutic and practical advantages in eligible cases of corneal trauma, particularly during a COVID-19 pandemic.

This has imposed new sanitary restrictions : limited access to the operating room in ophthalmology only for functional emergencies and a drastically reduced capacity for external consultations in favor of teleconsultation. The aim of this study is to evaluate the Vicryl 10-0 (polyglactin 910) resorbable monofilament suture in corneal trauma, rather than classic Nylon 10-0: structural and functional results, and adaptation of postoperative follow-up during a sanitary crisis period.

ELIGIBILITY:
Inclusion Criteria:

* Corneal penetrating injury and/or lamellar laceration

Exclusion Criteria:

* Corneal Penetrating injury trauma requiring necessarily ONLY Nylon 10-0
* Traumatism requiring necessarily a cryopreserved human amniotic membrane (for example)
* Traumatism eligible for biological glue (long-axis wound < 2 mm)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had an emergency eye surgery in the Saint-Etienne University Hospital from 18/03/2020 to 05/12/2020
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
change visual acuity (Snellen scale) from baseline and 2, 6, 12 and 18 months after the intervention | Months: 0, 2, 6, 12, 18
  Collected in the medical record.
change Visual acuity (Parinaud scale) from baseline and 2, 6, 12 and 18 months after the intervention | Months: 0, 2, 6, 12, 18
  Collected in the medical record.

SECONDARY OUTCOMES:
Astigmatism (diopter) | Months: 0, 2, 6, 12, 18
  Collected in the medical record. Measured by OCT-TOMEY-CASIA).
Number of postoperative external consultations | Months: 0, 2, 6, 12, 18
  Collected in the medical record.
Adverse events | Months: 0, 2, 6, 12, 18
  Collected in the medical record. All adverse events connecting to the eye surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Thibaut GARCIN, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No